CLINICAL TRIAL: NCT00802919
Title: Varenicline for Cognitive Deficits and Cigarette Smoking in Schizophrenia - Efficacy and Predictors, Independent Investigator Study
Brief Title: Varenicline for Cognitive Deficits and Cigarette Smoking in Schizophrenia - Efficacy and Predictors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Responsible Party: Principal Investigator, Robert C. Smith MD PhD, Research Psychiatrist, Principal Investigagtor, Nathan Kline Institute for Psychiatric Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 081/C02; FDA IND 102,411
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Schizophrenia; Cigarette Smoking
Keywords: schizophrenia; smoking; nicotine; cognitive deficits; nicotinic receptors; Cognitive Deficits in Schizophrenia
MeSH Terms: conditions — Schizophrenia; Cigarette Smoking; Smoking; Cognition Disorders | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline (Experimental): Varenciline 1-2 mg/day
  Interventions: Drug: Varenicline
- Matched Placebo (Placebo Comparator): placebo for varenicline
  Interventions: Drug: Placebo for varenicline

INTERVENTIONS:
Drug: Varenicline — Varenicline 1-2 mg/day
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo for varenicline — Placebo
  Arms: Matched Placebo

SUMMARY:
This is a 8-week double-blind placebo controlled parallel group study of the efficacy of varenicline (Chantix) for smoking cessation in schizophrenic patients, and its effect on cognitive function in patients with schizophrenia.At some sits evaluation of smoking measures is extended to 12 weeks. Correlations will be made with biological predictors of efficacy: a) measures of nicotinic receptors in lymphocytes b) DNMT1 and GAD67 mRNA in lymphocytes. Subjects will be current cigarette smokers or history of regular smokers.

DETAILED DESCRIPTION:
This was a double-blind placebo controlled study of varenicline and matched placebo in patients with a diagnosis of schizophrenia or schizoaffective psychosis who were treated with antipsychotic medication and were cigarette smokers. Three sites (2 U.S., 1 Israel) were supported by the Stanley grant. A similar independently supported study was conducted in Beijing, China. We were allowed to access these data and combine them for our analysis of results. Subjects at each site participated in a protocol which was approved by their institutional IRB. All subjects signed informed consent.

The study evaluated multiple measures of cigarette smoking, cognitive functions by MATRICS battery (Measurement and Treatment Research to Improve Cognition in Schizophrenia), and psychiatric symptoms by PANSS (Positive and Negative Symptom Scale), SANS (Schedule For Assessment Of Negative Symptoms), and Calgary Depression scales. Lymphocytes were collected for measurement of epigenetically related mRNA's.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Schizophrenia or Schizoaffective Disorder Current Cigarette Smoker or History of Chronic Cigarette smoking Age 18-65 Currently taking antipsychotic medication

Exclusion Criteria:

prior history of hospitalization for acute myocardial infarction or stroke, or persistent angina pectoris with current symptoms Patients who have previously tried varenicline and have stopped taking it because of side-effects of severe nausea or vomiting suicide attempt in the last year and or have had prominent or serious suicidal thoughts in the past year Women who are pregnant, nursing, or unable to use reliable contraception significant renal impairment(Creatinine ≥ 1.5) baseline Hamilton Depression Scores is >20

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2008-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Smith, MD, PhD, Principal Investigator — Nathan Kline Institute for Psychiatric Research
Locations (4):
- United States (2):
  - Manhattan Psychatirc Center, New York, New York
  - Nathan Kline Insitute for Psychiatric Research, Orangeburg, New York
- Peking University Institute of Mental Health, Beijing, China
- The Division of Psychiatry, Chaim Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Smith RC, Amiaz R, Si TM, Maayan L, Jin H, Boules S, Sershen H, Li C, Ren J, Liu Y, Youseff M, Lajtha A, Guidotti A, Weiser M, Davis JM. Varenicline Effects on Smoking, Cognition, and Psychiatric Symptoms in Schizophrenia: A Double-Blind Randomized Trial. PLoS One. 2016 Jan 5;11(1):e0143490. doi: 10.1371/journal.pone.0143490. eCollection 2016. PMID 26730716
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 93 subjects were consented, 2 withdrew consent before randomization, and 87 provided evaluable data on at least one outcome measure. The number enrolled 93, is less than the number started 91, because 2 patients withdrew consent before randomization
Period: Overall Study
Arm/Group | Varenicline | Matched Placebo
Started | 45 | 46
Completed | 42 | 45
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Matched Placebo | Total
Number analyzed (Participants) | 42 | 45 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (8.9) | 43.6 (10.6) | 44.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 35 | 39 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 14 | 13 | 27
  black-AA | 15 | 17 | 32
  hispanic | 5 | 7 | 12
  chinese han | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 22 | 27 | 49
  China | 8 | 8 | 16
  Israel | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Cotinine Level
Description: plasma cotinine
Time Frame: Baseline, 4 weeks, 8 weeks
Population: Data were available for cotinine analysis in mixed model analysis of co covariance on 34 participants in the varenicline arms and 36 participants in the placebo arm.
Measure: Mean (Standard Error); unit: cotinine ng/ml
Arm/Group | Varenicline | Matched Placebo
Number analyzed (Participants) | 34 | 36
cotinine ng/ml
  baseline | 257.9 (15.9) | 258.6 (18.4)
  week4 | 176.0 (16.0) | 252.1 (18.7)
  week8 | 147.0 (17.9) | 264.6 (18.9)

2. Primary Outcome: Change From Baseline in Cognitive Performance
Description: The MATRICS Consensus Cognitive Battery (MCCB)(Measurement and Treatment Research to Improve Cognition in Schizophrenia) was used to measure cognitive performance. Six Domain scores and a Composite score are calculated by the proprietary MCCB Computer Scoring Program (modified beta version) from raw scores on 10 individually administered subtests. The social cognition test was not assessed in this study. The Domain T-scores are percentile-ranked and range from <20 (<0.1 percentile) to >80 (>99.9 percentile). The Composite scores are also percentile-ranked and range from <213 (T<20, <0.1 percentile) to >487 (T>80, >99.9 percentile). Higher scores after baseline represent better outcomes. Here we report difference scores from post-treatment and baseline with positive difference scores representing better outcomes.
Time Frame: basline and 8 weeks (or end of study iif patient ended participation before the 8-weeks)
Population: N's varied from 25-32 in varenicline group and 29-35 in placebo group because all subjects did not complete all parts of MATRICS battery.Maximum number of participants is entered for number of participants because this cell entry does not allow entry of variable number of participations ( e.g. 25-32). for different scores..
Measure: Mean (Standard Error); unit: T scores from MATRICS battery
Arm/Group | Varenicline | Matched Placebo
Number analyzed (Participants) | 32 | 35
T scores from MATRICS battery
  MATRICS composite score diff from baseline: number analyzed (Participants) | 25 | 29
  MATRICS composite score diff from baseline | -0.19 (2.14) | 1.97 (1.86)
  MATRICS Speed of Processing diff from baseline: number analyzed (Participants) | 31 | 35
  MATRICS Speed of Processing diff from baseline | 3.03 (1.52) | 4.08 (1.56)
  MATRICS attention-vigilance diff from baseline: number analyzed (Participants) | 27 | 29
  MATRICS attention-vigilance diff from baseline | 2.49 (1.99) | 4.33 (1.95)
  MATRICS working memory diff from baseline | 0.95 (1.82) | 5.29 (1.88)
  MATRICS verbal learning diff from baseline | 0.94 (1.00) | 0.01 (1.04)
  MATRICS visual learning diff from baseline: number analyzed (Participants) | 31 | 35
  MATRICS visual learning diff from baseline | 4.75 (2.26) | 7.85 (2.30)
  MATRICS reasoning-rob sol diff from baseline: number analyzed (Participants) | 32 | 34
  MATRICS reasoning-rob sol diff from baseline | 0.38 (0.78) | 2.79 (0.81)

3. Secondary Outcome: Change From Baseline in Psychiatric Symptoms
Description: The Positive and Negative Syndrome Scale (PANSS) was used to measure psychiatric symptoms. Item scores ranged from 1 (Absent) to 6 (Severe) for symptoms on the Positive Scale (total subscale range: 7-42), the Negative Scale (total subscale range: 7-42), and the General Psychopathology Scale (total subscale range:16-96). All three subscales were summed for the PANSS total score (total scale range: 30-180). Scores closer to 30 after baseline represented better outcomes. Here we report difference scores from post-treatment and baseline with negative difference scores representing better outcomes.
Time Frame: baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Varenicline | Matched Placebo
Number analyzed (Participants) | 39 | 38
units on a scale
  PANSS Total wk4 -baseline diff | -3.56 (1.29) | -0.86 (1.42)
  PANSS Total wk8-baseline diff | -3.05 (1.35) | -0.97 (1.40)
  PANSS Depression Factor wk4-basline diff | -0.67 (0.24) | 0.23 (0.26)
  PANSS depressor factor wk8-baseline diff | -0.67 (0.25) | -0.10 (0.25)

4. Secondary Outcome: Change From Basellne in Calgary Depression Scale Score
Description: The Calgary Depression Scale for Schizophrenia. The scale has 9 items with ratings of 0 to 3 on each item. Total score can vary from 0 to 27. Higher scores indicate more depression. Negative change scores indicate decreasing depression.
Time Frame: baseline, 4 weeks, 8 weeks
Population: Not all patients had relevant responses on Calgary Depression Scale. Data are analyzed for 36 subjects randomized to varenicline and 38 subjects randomized to placebo (total N=74).
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Varenicline | Matched Placebo
Number analyzed (Participants) | 36 | 38
Scores on a scale
  Calgrapy Dep totl wk4-baseline diff | -0.63 (0.24) | -0.72 (0.27)
  calgrapy dep wk8-baseline diff | -0.79 (0.26) | -0.88 (0.26)

ADVERSE EVENTS:
Arm/Group | Varenicline | Matched Placebo
Serious Adverse Events (participants affected / at risk) | 2/45 | 1/46
Other Adverse Events (participants affected / at risk) | 0/45 | 0/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=45) | Matched Placebo (N=46)
psychiatric decompensation not study drug related (Psychiatric disorders) | 1 (1) | 0 (0) — after discharge from hospital patient decoenssated because of drug abuse and noncompliance with medication
auditory hallucination not study drug related (Psychiatric disorders) | 1 (1) | 0 (0) — patient developed auditory hallucinations although symptom scores had decreased on varenicline
verbal agression (Psychiatric disorders) | 0 (0) | 1 (1) — verbal aggression lead to [psychiatric hospitalization. Patient on placebo study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No